CLINICAL TRIAL: NCT07053410
Title: Comparison of Dimensional Accuracy and Color Stability Between Direct 3D-printed and Thermoformed Retainers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essraa hassan Hussein Mohamed (Other)
Responsible Party: Sponsor-Investigator, Essraa hassan Hussein Mohamed, Master's Degree Candidate in Orthodontics, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Orthodontic retainers
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Orthodontic Retention Appliance; Clear Orthodontic Retainers
Keywords: Direct 3D-printed retainers; Multilayer retainer; Singlelayer retainer

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel arms: 3D-printed retainers, single-layer thermoformed retainers, or multi-layer thermoformed retainers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T1 - 3D-Printed Retainers (Experimental): Participants in this group will receive retainers fabricated using direct 3D printing technology with bio-compatible clear resin.
  Interventions: Device: Direct 3D-Printed Retainer
- T2 - Single-Layer Thermoformed Retainers (Active Comparator): Retainers fabricated using thermoplastic sheets and a standard thermoforming machine.
  Interventions: Device: Single-Layer Thermoformed Retainer
- T3 - Multi-Layer Thermoformed Retainers (Active Comparator): Participants in this group will receive retainers fabricated using a multi-layer thermoforming method
  Interventions: Device: Multi-Layer Thermoformed Retainer

INTERVENTIONS:
Device: Direct 3D-Printed Retainer — Orthodontic retainers fabricated using direct 3D printing technology from digital STL models. The retainers are printed with biocompatible clear resin using an additive manufacturing process.
  Arms: T1 - 3D-Printed Retainers
Device: Single-Layer Thermoformed Retainer — Clear orthodontic retainers fabricated by thermoforming a single-layer thermoplastic sheet over a 3D printed dental model using a vacuum forming machine.
  Arms: T2 - Single-Layer Thermoformed Retainers
Device: Multi-Layer Thermoformed Retainer — Orthodontic retainers fabricated using a multi-layer thermoforming technique combining different thermoplastic materials to enhance durability and fit accuracy.
  Arms: T3 - Multi-Layer Thermoformed Retainers

SUMMARY:
This study aims to compare two types of orthodontic retainers used after active treatment to maintain teeth position. The retainers are fabricated using either direct 3D-printing or thermoforming methods. The study will evaluate which method provides better dimensional accuracy (fit) and color stability over time. Adult patients who have completed their orthodontic treatment will be randomly assigned to one of three groups, each receiving a different type of retainer. The research is conducted at the Faculty of Dental Medicine, Al-Azhar University - Assiut Branch. The goal is to help orthodontists select the most reliable and durable type of retainer for long-term use.

DETAILED DESCRIPTION:
This randomized clinical and laboratory study investigates the dimensional accuracy and color stability of orthodontic retainers fabricated using two different techniques: direct 3D printing and thermoforming. Patients who have completed active orthodontic treatment will be recruited and assigned to three groups. Group T1 will receive 3D-printed retainers, Group T2 will receive single-layer thermoformed retainers, and Group T3 will receive multi-layer thermoformed retainers…

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed their active orthodontic treatment.
* Adults aged 18 years and above.
* Cooperative individuals willing to participate.
* Patients with good oral hygiene and general health.
* No systemic diseases that may affect treatment outcomes.

Exclusion Criteria:

* Smokers.
* Patients with a history of poor compliance with previous orthodontic treatment.
* Patients with parafunctional oral habits (e.g., bruxism).
* Patients undergoing retreatment due to relapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mean Surface Deviation (mm) Between Retainer STL and Original STL Reference Model Assessed by 3D Superimposition After 1 Month | 1 month after retainer delivery
  Dimensional accuracy will be assessed by scanning each retainer and generating an STL file. The resulting STL will be superimposed on the original digital reference STL model using best-fit alignment in 3D inspection software (e.g., Geomagic Control X). The software will calculate the mean surface deviation in millimeters (mm). Results will be reported as mean ± standard deviation for each group (3D-printed vs thermoformed).

SECONDARY OUTCOMES:
Color Change (ΔE) of Retainers Measured by Spectrophotometer Based on CIE L*a*b* System After 1 Month | 1 month after retainer delivery
  Color stability will be evaluated by measuring the color of each retainer before and after intraoral use using a spectrophotometer. The color change (ΔE) will be calculated according to the CIE L*a*b* color system formula. Results will be reported as mean ΔE ± standard deviation for each group. A ΔE value >3.3 will be considered visually perceptible.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M. Dawaba, PhD, Principal Investigator — Faculty of Dental Medicine, Al-Azhar University - Assiut Branch
Locations (1):
- Faculty of Dental Medicine, Al-Azhar University - Assiut Branch, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No